CLINICAL TRIAL: NCT04039334
Title: The Effects of Creative Dance Based Exercise Training on Respiratory, Balance and Cognitive Functions, Respiratory and Peripheral Muscle Strength and Functional Capacity in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Meltem Kaya, Research Asistant, PT, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: bvumkaya01
Record Dates: First submitted 2019-07-26; First posted 2019-07-31 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: COPD
Keywords: COPD; Creative Dance; Exercise Training; 6 Minute Walk Test; Pulmonary Function Test; Postural Stability; Cognitive Functions; Muscle Strength
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Patients in this group will receive conventional chest physiotherapy, two times a day, 5 days a week for 8 week. All exercise sessions will be performed at home.
  Interventions: Other: Conventional Chest Physiotherapy
- Training Group (Experimental): In addition to conventional chest physiotherapy programme, patients in this group will also receive creative dance based exercise training for 60 minutes, 2 times in a week for 8 weeks. All exercise sessions will be supervised in a clinic per week.
  Interventions: Other: Conventional Chest Physiotherapy; Other: Creative Dance Based Exercise Training

INTERVENTIONS:
Other: Conventional Chest Physiotherapy — Conventional chest physiotherapy programme will include diaphragmatic breathing exercise, thoracic expansion exercises, incentive spirometer exercise (Triflo), teaching of respiratory control, relaxing and coughing techniques.
Other: Creative Dance Based Exercise Training — Creative dance based exercise training will be given under the supervision of a physiotherapist who takes creative dance instructor training 2 days and 60 minutes per week.
  Arms: Training Group

SUMMARY:
COPD is a common, preventable and treatable disease associated with an increased chronic inflammatory response of the airways and lungs to harmful gases and particles and characterized by progressive airflow restriction, which is usually progressive. Exercise intolerance is one of the most important outcomes of COPD. Dyspnea and leg fatigue are the main symptoms that limit exercise and patients restrict their activity to avoid these disturbing conditions. Exercise training is the most appropriate method for improving exercise tolerance and muscle function. It is considered and recommended by ERS and ATS as an essential component of PR. Endurance training is considered to be one of the most important components of the PR program. Walking, running, cycling, stair climbing, dancing are examples of endurance exercises. Dance-based exercise training; It is an entertaining method that increases physical, functional, cognitive, emotional and social integration. This alternative method has frequently been tried in the literature in the treatment of Parkinson's, cancer and psychiatric diseases and its effects on functional capacity, balance, and quality of life have been demonstrated. The importance of our research; This is the first study to apply dance based exercise training in chronic respiratory diseases.

The aim of this study was to investigate the effect of creative dance based exercise training on respiratory, balance and cognitive functions, respiratory and peripheral muscle strength and functional capacity in COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Having FEV1 / FVC <70% from pulmonary function test
* Being older than 18 years
* To be able to read and understand Turkish

Exclusion Criteria:

* No exacerbation in 8 weeks.
* Attending current or regular exercise training in the last 1 year
* Having diagnosed vision, hearing, vestibular or neurological problems that may affect balance
* Having orthopedic, musculoskeletal or cardiovascular comorbid conditions that may affect ambulation
* Being on long-term oxygen therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Respiratory Function Test | Eight weeks
  Change from baseline forced vital capacity (FVC) at 8 weeks.
Respiratory Function Test | Eight weeks
  Change from baseline forced forced expiratory volume in 1 second at 8 weeks.
Respiratory Function Test | Eight weeks
  Change from baseline peak expiratory flow (PEF) at 8 weeks.
COPD Assessment Test (CAT) | Eight weeks
  Change from baseline CAT score at 8 weeks.
BODE Index | Eight weeks
  Change from baseline BODE score at 8 weeks.
Balance | Eight weeks
  Change from baseline postural stability test score in BIODEX Balance System at 8 weeks.
Balance | Eight weeks
  Change from baseline limits of stability test score in BIODEX Balance System at 8 weeks.
Respiratory Muscle Strength | Eight weeks
  Change from baseline maximum inspiratory pressure at 8 weeks.
Respiratory Function Test | Eight weeks
  Change from baseline maximum expiratory pressure at 8 weeks.
Functional Capacity | Eight weeks
  Change from baseline distance covered in six minute walk test at 8 weeks.
Change from baseline handgrip strength at 8 weeks. | Eight weeks
  Change from baseline m. quadriceps strength at 8 weeks.
Change from baseline handgrip strength at 8 weeks. | Eight weeks
  Change from baseline m. biceps strength at 8 weeks.
Change from baseline handgrip strength at 8 weeks. | Eight weeks
  Change from baseline handgrip strength at 8 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Department of Physiotheraphy and Rehabilitation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided